CLINICAL TRIAL: NCT06875739
Title: An Innovative Method in SAliva Samples for the Early Differential Diagnosis of High-impact NeuroDegenerative Diseases Through Raman Spectroscopy
Acronym: SANDY
Status: Enrolling by invitation | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: University of Cagliari, Cagliari, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: SANDY - POC
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-10

CONDITIONS: Neurodegenerative Disorders; Parkinson Disease; Alzheimer Disease; Parkinsonian Disorders; Fronto-temporal Dementia; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Neurodegenerative Diseases; Parkinson Disease; Alzheimer Disease; Parkinsonian Disorders; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control subjects: They are subjects admitted to IRCCS Don Gnocchi Florence in the cardiology, pulmonology, and orthopedics departments who have no neurological symptoms or diagnosis of neurological or psychiatric diseases, in the absence of positive family history (relatives I and II degree) for NDDs. Control subjects should be in a clinically stable condition at inclusion, and will be enrolled at least 15 days after the acute event causing hospitalization.
- cases: They are individuals with a diagnosis of alzheimer's dementia, diagnosis of fronto-temporal dementia(behavioral variant), diagnosis of Parkinson's disease, clinical diagnosis of Parkinsonisms, and clinical diagnosis of amyotrophic lateral sclerosis.
- prodromal cases: Subjects with Parkinson's or Alzheimer's disease or Frontotemporal dementia (behavioral variant) in the prodromal stage according to Berg's criteria.

SUMMARY:
The aim of the study is to validate a salivary test that allows for rapid and accurate objective diagnosis in the context of neurodegenerative diseases, a complex of diseases that includes Alzheimer's Dementia, Frontotemporal Dementia, Parkinson's Disease, Atypical Parkinsonisms, and Amyotrophic Lateral Sclerosis. In particular, the study aims to validate the salivary method against methods already in use (CSF method) or better studied (blood-based method) to allow early recognition of the disease condition and a distinction between the various diseases in order to receive appropriate therapy when possible.

In fact, the term neurodegenerative diseases is a broad term that includes disorders characterized by predominantly cognitive, motor, or mixed disorders for which early and accurate diagnosis of the disease is often difficult given also the variability with which these diseases can present. Ab initio recognition of a specific neurodegenerative disease would allow better pharmacological management of this disorder and facilitate the planning of care and rehabilitation interventions. In general, the recognition of neurodegenerative diseases could be facilitated by the use of a biomarker, which is a biological indicator that can be related to the onset or development of a disease. For this reason, it is necessary to compare the biomarker assay of patients with that of controls, so you were asked to participate as a "Control Subject" precisely because you do not have neurodegenerative disease.

Participation in the study involves, in addition to the collection of clinical-demographic data, the performance of a cognitive screening test to attest that your cognitive performance is in the normal range and the collection of biological blood and salivary samples, to be compared with those of participants with neurodegenerative diseases. Apolipoprotein E (ApoE) polymorphism study will be performed on the blood. A genetic polymorphism is a variation in the DNA sequence present in at least 1% of the population, the determination of ApoE polymorphism will allow to define a His genetic characteristic related to a higher or lower risk of developing Alzheimer's Disease. Two specific biomarkers, called neurofilament light chain (NfL) and gliofibrillary acidic protein (GFAP), namely a marker of neurodegeneration and one of neuroinflammation, will also be assayed on blood. Analysis of some inflammatory proteins called cytokines will also be performed.

On saliva, the biochemical composition will be evaluated with the analysis of particles present within it called vesicles by a method called Raman Spectroscopy, and the assay of specific biomarkers called NfL and GFAP will also be performed on saliva. The diagnosis of pathology made according to clinical diagnostic criteria and supported, when necessary, by the presence of recognized biomarkers (molecular imaging/liquid markers) will be used as a reference to evaluate the diagnostic capabilities of salivary methodology to detect different pathologies and to differentiate a pathological condition from Controls. Finally, the study will also include a comparison of salivary study methods on a group of people who are at a very early stage of disease, in order to detect whether the study performed with portable instrumentation is as good a method as that with laboratory instrumentation. In fact, the use of portable instrumentation would make it even easier to acquire a biomarker quickly directly from the clinic.

ELIGIBILITY:
Inclusion Criteria:

FOR ALL SUBJECTS: between 60 and 85 years old

FOR CASE:

1. ADD: diagnosis of dementia due to AD according to clinical criteria and supported by amyloid biomarkers (biomarkers in CSF or brain PET scan with amyloid-specific tracer) according to the definition biological or neurochemical definition of disease.
2. FTD: diagnosis of FTD-bv (behavioral variant) according to current clinical criteria.
3. PD: diagnosis according to MDS criteria; stable drug treatment (last 4 weeks).
4. APs: clinical diagnosis of Progressive Supranuclear Palsy according to the criteria of Hoglinger 2017, Corticobasal Degeneration according to the criteria of Armostrong 2013, Multisystem Atrophy according to the criteria of Wenning 2022.
5. ALS: clinical diagnosis according to the criteria of Brooks (2000) and subsequent revisions.

FOR CONTROL SUBJECTS

1. subjects admitted to IRCCS Don Gnocchi Florence in the departments of cardiology, pulmonology, orthopedics
2. ABSENCE of neurological symptoms
3. ABSENCE OF diagnosis of neurological or psychiatric diseases.
4. absence of positive family history (relatives I and II degree) for NDDs.
5. condition of clinical stability
6. at least 15 days after the acute event causing hospitalization.

FOR PRODROMAL CASE

1. Prodromal PD according to Berg's criteria.
2. prodromal FTD-bv according to Barker's criteria
3. prodromal AD according to the criteria of Dubois and Albert

Exclusion Criteria:

FOR CASE

1. Vascular Parkinsonism and other forms of secondary Parkinsonism such as drug-induced, other known or suspected causes (metabolic, brain tumor, etc.).
2. MoCA<15 for subjects with PD
3. cases with validated biomarkers (CSF and PET) in diagnostic conflict.

FOR ALL SUBJECTS

1. significant comorbidities
2. presence of severe systemic diseases or previously diagnosed psychiatric illnesses
3. patients unable to express consent for participation in the study themselves
4. presence of clinically unstable oral cavity disease (inflammatory/infectious)
5. time since acute event (if it occurred) <15 days
6. presence of local or systemic infection/inflammation detected on routine examinations.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NDDs will be recruited from participating centers through enrollment. We plan to recruit at least 52 subjects per experimental group (52 ADDs, 52 FTDs, 52 PDs, 52 APs, 52 ALS) and 50 CTRLs. An additional 50 prodromal cases belonging to the PD, FTD behavioral variant, and AD categories.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative Illness Rating Scale (CIRS) | at enrollment
  it's a scale that records the comorbidity
Neurological Clinical informations | at enrollment
  Presence/absence of symptoms/signs such as presence of speech disorder, hearing loss, low vision, dysphagia, oculomotricity disorder, disorientation, decreased insight, fatuity, perseveration/affacceleration, dx/sn recognition inability, gait disorder, instability/falls, neglect, ideomotor apraxia, signs of frontal release, rigidity/spasticity, bradykinesia, tremor or other involuntary movements, signs of first or second motor neuron, need for use of aids/presence of medical aids.
Genetic test | at enrollment
  genetic testing will lead in NDDs and CTRL to the determination of the ApoE polymorphism (categorical variable). In NDDs, diagnostic investigation will aim to confirm/exclude a mutation in one of the disease-causing genes (APP, PS1, PS2, MAPT, PGRN, C9ORF72, SOD 1, TARDBP, VCP) in accordance with the pathological phenotype
Plasma test | at enrollment
  NfL and GFAP assay result on plasma (continuous numeric variables)
Salivary test | at enrollment
  results of NfL and GFAP assay on saliva (continuous numeric variables)
nerological objective examination checklist | at enrollment
  presence/absence of symptoms/signs such as presence of speech disorder, hearing impairment, low vision, dysphagia, oculomotor disorder, disorientation, decreased insight, fatuity, perseveration/affacility, dx/sn recognition inability, gait disorder, instability/falls, neglect, ideomotor apraxia, signs of frontal release, rigidity/spasticity, bradykinesia, tremor or other involuntary movements, signs of first or second motor neuron,need for use of aids/presence of medical aids (categorical variables)
UPDRS part III and IV | at enrollment
  evaluation of motor symptoms only for subjects with parkinson's disease or parkinsonisms
Hoehn and Yahr Scale | at enrollment
  evaluation of clinical status only for subjects with parkinson's disease
NON-MOTOR SYMPTOMS SCALE | at enrollment
  evaluation of non motor symptoms only for subjects with parkinson's disease
Functional Rating Scale-Revised (ALSFRS-R) | at enrollment
  evaluation of disability only for subjects with ALS
MONTREAL COGNITIVE ASSESSMENT (MOCA) | at enrollment
  Cognitive screening test for all except control subjects
denomination test of SAND | at enrollment
  denomination of visual stimuli for all subjects except control cases
semantic, phonemic and alternate fluency Test | at enrollment
  semantic, phonemic and alternate fluency Test for all subjects except control cases
TRAIL MAKING TEST part A and B | at enrollment
  evaluation of attentional skills for all subjects except control cases
STROOP TEST | at enrollment
  evaluation of inhibitory control for all subjects except control cases
REY'S 15-WORD TEST | at enrollment
  evaluation of long term memory for all subjects except control cases
REY OSTERRIETH COMPLEX FIGURE | at enrollment
  evaluation of visuospatial skills for all subjects except control cases
FACE TEST | at enrollment
  evaluation of ability to recognize mental states of others for all subjects except control cases
NEUROPSYCHIATRICH INVENTORY (NPI) | at enrollment
  interview assessing behavioral of others for all subjects except control cases
FRONTAL ASSESSMENT BATTERY (FAB) | at enrollment
  evaluation of executive functions; for all subjects except control cases
MINIMENTAL STATE EXAMINATION (MMSE) | at enrollment
  cognitive screening only for subjects with ADD and with Mild Cognitive Impairment (MCI)

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Azienda Ospedaliera Universitaria di Cagliari, Cagliari
  - IRCCS Fondazione Don Carlo Gnocchi, Florence
  - Laboratorio Congiunto di Ricerca DON GNOCCHI - UNIFI neurogenetica in riabilitazione - NGR, Florence
  - IRCCS Fondazione Don Carlo Gnocchi, Milano, Milan